CLINICAL TRIAL: NCT02170649
Title: The Tolerability and Effect of Food on the Pharmacokinetics of a Single 800 mg Oral Dose of BIA 2-093 in Healthy Male Volunteers
Brief Title: The Tolerability and Effect of Food on the Pharmacokinetics of a Single 800 mg Oral Dose of BIA 2-093
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-103
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-03

CONDITIONS: Epilepsy
Keywords: BIA 2-093; Eslicarbazepine acetate
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group (Experimental): the volunteers received a single 800 mg BIA 2-093 following either a standard high fat content breakfast or 10 hours of fasting. Fed and fasting periods were separated by a washout period
  Interventions: Drug: BIA 2-093

INTERVENTIONS:
Drug: BIA 2-093
  Other Names: ESL, Eslicarbazepine acetate

SUMMARY:
The purpose of this study is to investigate the effect of food on the pharmacokinetics of a single 800 mg oral dose of BIA 2-093 in healthy volunteers.

DETAILED DESCRIPTION:
Single centre, open label, randomized, two-way crossover study in 12 healthy male volunteers. The study consisted of 2 periods separated by a washout period of 14 days or more. On each of the study periods the volunteers received a single 800 mg oral dose of BIA 2-093 following either a standard high fat content breakfast or 10 hours of fasting.

ELIGIBILITY:
Inclusion Criteria:

Subjects were eligible for entry into the study if they fulfilled the following inclusion criteria:

* Male subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 28 kg/m2, inclusive.
* Subjects who were healthy as determined by pre study medical history, physical examination, neurological examination, EEG, and 12-lead ECG.
* Subjects who had clinical laboratory tests clinically acceptable to the investigator.
* Subjects who were negative for HBsAg, anti-HCV Ab and HIV-1 and HIV-2 Ab tests at screening.
* Subjects who were negative for alcohol and drugs of abuse at screening and admission.
* Subjects who were non-smokers or who smoked less than 10 cigarettes or equivalent per day.
* Subjects who were able and willing to give written informed consent.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria.
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 21 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening and/or admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening and/or admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Subjects who had an acute infection such as influenza at the time of screening and/or admission.
* Subjects who had used prescription drugs within four weeks of first dosing.
* Subjects who had used over-the-counter medication excluding oral routine vitamins but including mega dose vitamin therapy within one week of first dosing.
* Subjects who had used any investigational drug and/or participated in any clinical trial within two months of their first admission to this study.
* Subjects who had previously received BIA 2-093.
* Subjects who had donated and/or received any blood or blood products within the previous two months prior to screening.
* Subjects who were vegetarians, vegans and/or had medical dietary restrictions.
* Subjects who could not communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2001-09; Primary Completion 2001-11 (Actual); Study Completion 2001-11 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- BIA 2-093 (Fasting & Fed): 2 periods separated by a washout period of 14 days or more, on each of the study periods the volunteers received a single 800 mg oral dose of BIA 2-093 following either a standard high fat content breakfast or 10 hours of fasting.
Period: Fasting Period
Arm/Group | BIA 2-093 (Fasting & Fed)
Started | 12
Completed | 12
Not Completed | 0
Period: Fed Period
Arm/Group | BIA 2-093 (Fasting & Fed)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Fasting Period: single 800 mg oral dose of BIA 2-093 following 10 hours of fasting or following either a standard high fat content breakfast.
Arm/Group | Fasting Period
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Maximum observed plasma concentration of BIA 2-093
Time Frame: pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72 and 96 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Single Group: 2 periods separated by a washout period of 14 days or more, on each of the study periods the volunteers received a single 800 mg oral dose of BIA 2-093 following either a standard high fat content breakfast or 10 hours of fasting.
Arm/Group | Single Group
Number analyzed (Participants) | 12
ng/mL
  Fasting | 11302 (1866)
  Fed | 12799 (1769)

2. Secondary Outcome: Time of Occurrence of Cmax (Tmax)
Description: Time of occurrence of Cmax of BIA 2-093
Time Frame: pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72 and 96 hours post-dose
Measure: Median (Full Range); unit: hours
Arm/Group | Single Group
Number analyzed (Participants) | 12
hours
  Fasting | 3.5 [0.5 to 8.0]
  Fed | 4.0 [0.5 to 8.0]

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Sampling Time at Which Concentrations Were at or Above the Limit of Quantification (AUC0-t)
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time at which concentrations were at or above the limit of quantification (AUC0-t) of BIA 2-093
Time Frame: pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72 and 96 hours post-dose
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Single Group
Number analyzed (Participants) | 12
ng.h/mL
  Fasting | 243155 (31213)
  Fed | 229350 (41366)

4. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity (AUC0-oo)
Description: Area under the plasma concentration versus time curve from time zero to infinity (AUC0-oo) of BIA 2-093
Time Frame: pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, 72 and 96 hours post-dose
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Single Group
Number analyzed (Participants) | 12
ng.h/mL
  Fasting | 243589 (31052)
  Fed | 242459 (32085)

ADVERSE EVENTS:
Arm/Group | Single Group
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 10/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Group (N=12)
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 1
Gastroenteritis NOS (Infections and infestations) | 1
Rhinosinusitis (Infections and infestations) | 1
Headache NOS (Nervous system disorders) | 2
Muscle contraction involuntary (Nervous system disorders) | 1
Nystagmus (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1
Myalgia of lower extremities (Musculoskeletal and connective tissue disorders) | 1
Dry cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis NOS (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus NOS (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other